CLINICAL TRIAL: NCT04269798
Title: The Effect of Functional Electrical Stimulation Technology on Gait and Balance Performance in Children With Hemiplegic Cerebral Palsy
Brief Title: The Effect of Functional Electrical Stimulation on Gait and Balance in Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Shamekh Mohamed El-Shamy, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Umm AlQura University
Record Dates: First submitted 2020-02-09; First posted 2020-02-17 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Treatment Arm (Active Comparator): Will receive conventional rehabilitation program for the lower limbs, balance and gait training. Two hours of conventional physical therapy program /session - 3 sessions/week/ three successive months.
  Interventions: Other: Traditional Treatment
- Functional Electrical Stimulation Group (Experimental): Will receive 1.5 hours of conventional physical therapy program /session - 3 sessions weekly - three successive months + 1/2 hour of the gait training program with functional electrical stimulation /session - 3 sessions weekly - three successive months.
  Interventions: Other: Traditional Treatment

INTERVENTIONS:
Other: Traditional Treatment — conventional rehabilitation program for lower limb, balance and gait training

SUMMARY:
The aim of this study will be to evaluate the effect of FES on stimulation of the anterior tibial group by using the WalkAide foot drop stimulator on improving walking and balance abilities in children with hemiplegic CP.

DETAILED DESCRIPTION:
The aim of this study will be to evaluate the effect of FES on improving walking and balance abilities in children with hemiplegic CP. Forty children with hemiplegic CP will be assigned randomly into two groups (A & B). Control group (A) will receive conventional rehabilitation program for lower limb, balance and gait training. Study group (B) will receive conventional rehabilitation program as in group (A) in addition to FES by using the WalkAide foot drop stimulator. Patients' evaluation will be carried out before and after training to assess walking ability and balance performance.

ELIGIBILITY:
Inclusion Criteria:

* Their weight should be less than 40 kg.
* The spasticity degrees of the affected lower limb will range between grades (1, 1+ & 2) according to Modified Ashworth Scale (MAS).

Those children functioning scores at Gross Motor Function Classiﬁcation System (GMFCS) Levels I and II.

* They can walk 10 min conditionally without an orthosis.
* Ought to be intellectually skilled and ready to comprehend and take after directions.
* They will have neither serious nor recurring medical complications.
* Children's height will be more than 100 cm to fit with the Biodex balance equipment that will be used in this study to evaluate balance performance.
* No serious hip & knee flexion tightness will be present. Knee flexion at starting contact should be between 20-40º .
* Peroneal nerve and the proximal leg muscles ought to be in place.
* They ought to have no significant issues influencing balance other than spasticity.

Exclusion Criteria:

* Children who demonstrate skin diseases or allergic reactions to adhesive tape or any other materials used in this study.
* Children with visual, auditory or perceptual deficits.
* Children with surgical interference for the lower limb.
* Children with seizures or epilepsy.
* Children who received botulinum toxin in the lower extremity musculature during the past 6 months or who wish to receive it within the period of study, other spasticity medication within 3 months of pre-treatment testing .
* Children with pacemakers or other diseases that are contraindicated by electrical stimulation.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline spatial and temporal gait analysis at 3 months | Baseline and 3 months post-intervention
  Spatial and temporal gait analysis will be evaluated for every child at baseline and 3 months post-intervention using the Noraxon's Myo PRESSURE plate.
Change from baseline postural stability at 3 months | Baseline and 3 months post-intervention
  Postural stability will be evaluated at baseline and 3 months post-intervention using the Biodex Balance System (BBS) (Balance System SD, Shirely, NY, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Shamekh M El-Shamy, Ph.D., Principal Investigator — Professor
Locations (1):
- Maternity and Children Hospital, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No